CLINICAL TRIAL: NCT06899256
Title: The Effect of Horticultural Activities on Physical and Cognitive Status, Mental Well-Being, Social Participation and Quality of Life in Individuals Diagnosed with Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Betul Ustün, Occupational therapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10470346
Record Dates: First submitted 2024-11-14; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Dementia; Horticultural Therapy; Quality of Life; Occupational Therapy; ELDERLY PEOPLE
Keywords: dementia; horticultural activity; nursing homes; quality of life
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): This horticultural activity program was not implemented.
- Intervention Group (Experimental): This horticultural activity program was implemented.
  Interventions: Other: Horticultural Activity Program

INTERVENTIONS:
Other: Horticultural Activity Program — Prior to the commencement of the horticultural intervention program, the nursing home was visited to assess its physical environment and to inform staff about the program's objectives. Participants were recruited, and baseline data was collected. The program was structured around weekly activities and visits, with a three-day interval between each session. Activities included plant identification, gardening tasks, and nature-based art projects. The program was designed to foster social interaction, cognitive stimulation, and physical activity, while promoting a sense of accomplishment and well-being among participants. Throughout the program, regular assessments were conducted to monitor participants' progress and satisfaction.
  Arms: Intervention Group

SUMMARY:
This study aims to examine the effects of horticultural activities on the physical and cognitive status, mental well-being, social participation, and quality of life of individuals diagnosed with dementia living in nursing homes. Forty individuals participated in the study. The intervention group received a 10-week horticultural activity program, conducted two days a week (one activity day and one visit day), while the control group underwent evaluations without participating in the horticultural activities. Various standardized assessment tools were used to evaluate mental status, functional mobility, cognitive performance, mental well-being, social participation, and quality of life.

DETAILED DESCRIPTION:
The objective of this study is to investigate the impact of a structured horticultural activity program on individuals diagnosed with dementia who reside in nursing homes. The study was conducted with a total of 40 participants. The intervention group participated in a 10-week horticultural activity program, held twice weekly, which included one activity session and one visit session per week. The control group did not participate in the activity program but underwent the same evaluation procedures.

The assessment tools used in this study included:

Mini Mental State Examination to evaluate mental status, Timed Up and Go Test to assess functional mobility, balance, and performance, Rapid Mild Cognitive Impairment Test for cognitive assessment, Warwick-Edinburgh Mental Well-Being Scale to measure mental well-being, Social and Emotional Loneliness Scale for Adults to assess social and emotional loneliness, World Health Organization Quality of Life Scale Elderly Module to evaluate quality of life.

The study is designed to explore whether horticultural activities can be beneficial as part of occupational therapy interventions for individuals with dementia living in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

Residents of a nursing home Age 65 years or older Diagnosed with dementia Mini Mental State Examination (MMSE) score of 18 or higher

Exclusion Criteria:

Orthopedic dependency requiring the use of a wheelchair Diagnosed with any neurological or psychological disorder other than dementia

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Mini Mental State Examination Score | Baseline and Week 10
  Assessment of participants' cognitive status using the Mini Mental State Examination (MMSE). Scores will be recorded at baseline and after the 10-week intervention period.
Timed Up and Go Test Performance | Baseline and Week 10
  Evaluation of participants' functional mobility, balance, and performance using the Timed Up and Go Test. Results will be recorded at baseline and after the 10-week intervention period.
Rapid Mild Cognitive Impairment Test Score | Baseline and Week 10
  Assessment of cognitive status using the Rapid Mild Cognitive Impairment Test. Scores will be recorded at baseline and after the 10-week intervention period.
Warwick-Edinburgh Mental Well-Being Scale Score | Baseline and Week 10
  Measurement of mental well-being using the Warwick-Edinburgh Mental Well-Being Scale. Scores will be recorded at baseline and after the 10-week intervention period.
Social and Emotional Loneliness Scale for Adults Score | Baseline and Week 10
  Assessment of social and emotional loneliness using the Social and Emotional Loneliness Scale for Adults. Scores will be recorded at baseline and after the 10-week intervention period.
World Health Organization Quality of Life Scale Elderly Module Score | Baseline and Week 10
  Evaluation of participants' quality of life using the WHOQOL-OLD scale. Scores will be recorded at baseline and after the 10-week intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Betül Üstün, Merkez, Isparta, Turkey (Türkiye)